CLINICAL TRIAL: NCT03335306
Title: Epidemiological Study on Body Constitution Classified by Traditional Chinese Medicine Theory
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Wendy Wong, Professor, Chinese University of Hong Kong
Other Study IDs: HKCTR-1355
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Body Constitution
Keywords: Body constitution; Chinese Medicine; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy subjects in Hong Kong

SUMMARY:
Background: Different people are classified into different physiological constitution types in the Traditional Chinese Medicine (TCM) theory. Two instruments, the Body Constitution Questionnaire (BCQ) and the Constitution in Chinese Medicine Questionnaire (CCMQ), have been developed in Taiwan and Mainland China respectively to measure constitution. They were adapted and pilot tested in primary care Chinese patients in Hong Kong, which showed acceptable validity and reliability. These instruments have potential applications for epidemiological studies on body constitution.

Aim and objectives: The aim of this study is to establish the prevalence and epidemiology of body constitution classified by the Traditional Chinese Medicine Theory in the Chinese population in Hong Kong. It would also determine whether the prevalence of constitution types change with seasons and whether it is associated with socio-demographic factors, place of origin or residence, life style, or quality of life.

Design and subjects: Two cross-sectional telephone surveys of the Hong Kong (HK) general Chinese population, one in Summer and one in Winter, will be carried out. Sample size for each survey is 3200 subjects.

Methods: Residential-telephone-owning households will be contacted through random dialing by the Social Science and Research Centre of the University of Hong Kong using the Computer-Assisted Telephone Interviewing (CATI) system that covers 95% households in Hong Kong. A member, aged 18 or above, of the contacted household who last had his/her birthday will be invited to the study to answer either the BCQ or the CCMQ and a structured questionnaire on socio-demographics, place of origin, place of residence, health service utilization, life style and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Can be contacted by in a residential telephone number
* Age 18 or above
* Chinese who can communicate in Cantonese or Chinese by telephone;
* Has given verbal consent to take part in the study

Exclusion Criteria:

* Cannot communicate in Cantonese or Chinese
* Persons who cannot communicate by telephone;
* Refuse to give consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Methods: Residential-telephone-owning households will be contacted through random dialing by the Social Science and Research Centre of the University of Hong Kong using the CATI system that covers 95% households in Hong Kong. A member, aged 18 or above, of the contacted household who last had his/her birthday will be invited to the study to answer either the BCQ or the CCMQ and a structured questionnaire on socio-demographics, place of origin, place of residence, health service utilization, life style and quality of life.
Sampling Method: Probability Sample
Enrollment: 6400 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of constitution types classified by the BCQ or CCMQ | Baseline only
  Proportion of different constitution types according to the BCQ or CCMQ questionnaire

SECONDARY OUTCOMES:
Short Form-12 (SF-12) Health-related quality of life of people with different constitution types | Baseline only
Chinese quality of life (ChQOL) (HK version) Health-related quality of life of people with different constitution types | Baseline only

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hksar, China